CLINICAL TRIAL: NCT00695240
Title: Post-Operative Pain Control Using Direct Continuous Bupivacaine Infusion After Pelvic Organ Prolapse Repair
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Kansas City, Missouri (Other)
Responsible Party: Marilyn Horn, Institutional Review Board
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-310
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Post-Operative Pain; Pelvic Organ Prolapse
Keywords: Continuous bupivacaine infusion; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Pelvic Organ Prolapse; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bupiv analgesia (Experimental): Patients assigned to the study group had an ON-Q PainBuster Post-Op Pain Relief System (270 ml x 4 ml/hr, dual catheter, 2 ml per site, 72 hours continuous) with dual five inch fenestrated catheters placed at the sacrospinous ligament. The catheter was placed in the operating room with a peel-away trocar and attached to the pump. The trocar was inserted through a 5 mm stab incision made near the superior part of the pubic bone between the genitoinguinal fold and the midline of the symphysis. Once through the incision, the trocar is advanced subcutaneously and made to exit the posterior fourchette just beneath the posterior vaginal mucosa where it is advanced by tenting up the skin.
  Interventions: Device: Continuous bupivacaine analgesia infusion (ON-Q PainBuster Post-Op Pain Relief System)

INTERVENTIONS:
Device: Continuous bupivacaine analgesia infusion (ON-Q PainBuster Post-Op Pain Relief System) — Patients assigned to the study group had an ON-Q PainBuster Post-Op Pain Relief System (270 ml x 4 ml/hr, dual catheter, 2 ml per site, 72 hours continuous) with dual five inch fenestrated catheters placed at the sacrospinous ligament. One half percent bupivacaine was utilized.
  Other Names: ON-Q PainBuster Post-Op Pain Relief System

SUMMARY:
This prospective randomized controlled study will determine the efficacy of continuous local anesthesia at decreasing pain scores compared to patient controlled analgesia for pelvic organ prolapse procedures including posterior colporrhaphy and sacrospinous ligament fixation.

DETAILED DESCRIPTION:
Direct post-operative analgesia can be administered via a direct continuous analgesia pumps providing local anesthetic into a dissected area. To date, no studies have been conducted to evaluate pain control or infection with vaginal placement of catheters for pelvic organ prolapse surgery. To help pelvic surgeons assess the relative benefit of continuous local infusion of topical anesthetic following sacrospinous ligament fixation versus PCA pump, we compared pain scores, narcotic, anti-pruritic and anti-emetic drug usage, and wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Female patients greater than 18 years of age
* Undergoing posterior colporrhaphy at Saint Lukes Hospital, Kansas City, MO.

Exclusion Criteria:

* Patients with chronic pain conditions requiring daily narcotics were excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was a difference in the Wisconsin Brief Pain Inventory and Visual Acuity Score after treatment with the direct continuous analgesia device compared to PCA alone. | Each day post-operatively

SECONDARY OUTCOMES:
Secondary outcome was differences in the amount of narcotics, NSAIDS, antiemetics, time to return of bladder function, and complications between the study groups. | Each day post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Tyler M Muffly, MD, Study Director — St. Luke's Hospital
Locations (1):
- St. Luke's Hospital, Kansas City, Missouri, United States